CLINICAL TRIAL: NCT06601439
Title: Utilization of Maternal Healthcare Services and Infant Feeding Practices Among Slum-Dwelling Women in Pune, India
Brief Title: Utilization of Maternal Healthcare Services and Infant Feeding Practices
Acronym: HTHMCH
Status: Active, not recruiting | Type: Observational
Sponsor: Hirabai Cowasji Jehangir Medical Research Institute (Other)
Responsible Party: Principal Investigator, Dr. Anuradha Khadilkar, Deputy Director, Hirabai Cowasji Jehangir Medical Research Institute
Other Study IDs: JCDC/BHR/24/045
Record Dates: First submitted 2024-07-16; First posted 2024-09-19 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Maternal Health; Prenatal Care; Feeding Patterns
MeSH Terms: conditions — Feeding Behavior | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Observational Study — Observational Study

SUMMARY:
The goal of this observational study is to assess household food insecurity among slum-dwelling women in India and to explore if household food insecurity is associated with maternal healthcare services utilization and infant feeding practices

The main questions it aims to answer are:

1. Is the utilization of maternal healthcare services antenatally, during delivery, and postnatally associated with household food insecurity among slum-dwelling women in Pune, India?
2. Is household food insecurity associated with birth outcomes and infant growth in these women?

Participants will be asked:

1. For information related to socio-demographic characteristics, healthcare services utilization, food insecurity experience, dietary intake, and infant feeding indicators using a questionnaire.
2. Anthropometric measurements of the participant, her husband and her infant/s will be collected.
3. Focus group discussions (FGDs) will also be conducted to gain insight into the perceptions of these women with respect to the utilization of maternal healthcare services.

DETAILED DESCRIPTION:
The first target indicator of Sustainable Development Goal (SDG) 3 i.e. Good Health and Well-being for all at all ages is reducing the global maternal mortality ratio (MMR) to less than 70 per 100,000 live births by 2030. India, however, has been performing well on this indicator with progressive reduction in MMR from 130 deaths per 100,000 live births in 2014-16 to 97 deaths per 100,000 live births in 2018-2020, with eight Indian states achieving the SDG target of MMR to less than 70, where Maharashtra ranks 2nd amongst these states. It is well-known that the appropriate utilization of maternal healthcare services contributes to reduced maternal morbidity and mortality and improved offspring health. Women who availed of even one antenatal care (ANC) visit were more likely to opt for institutional deliveries and postnatal care. India provides comprehensive continuum of care in maternal and newborn health comprising quality ANC, delivery care, and postnatal care (PNC). However, there is considerable regional inequity in the utilization of these services. There are multiple factors that influence the utilization of maternal healthcare services which vary by region, religion, socio-economic status, and service delivery environment among many others. Thus, it is imperative to identify enablers, barriers and need gaps location wise so that appropriate interventions can be developed for promotion of healthcare service utilization. Pune has been reported to have an MMR of 49 per 100,000 live births, however, there are limited data on MMR among slum-dwelling women. Also, there are inadequate data on maternal healthcare utilization among slum-dwelling women in Pune. Given that need gaps in the continuum of care for maternal healthcare services are unique to socio-economic status and location, it is important to conduct a needs assessment for utilization of maternal healthcare services among slum-dwelling women in Pune. Moreover, as care in the antenatal period is linked not only to improved maternal health but also to newborn and infant survival and health, it is important to assess birth outcomes and infant growth in relation to maternal utilization of healthcare services. Food insecurity negatively impacts pregnant and lactating women as gender biases may interfere with their access to adequate food thus, affecting their health and the health of their offspring. Thus, it was deemed necessary to assess household food insecurity among slum-dwelling pregnant women in India and to explore if household food insecurity is associated with maternal healthcare services utilization.

Therefore, this study has been planned with the following objectives:

1. To assess the utilization of antenatal and postnatal health care services by slum-dwelling women from Pune
2. To assess infant feeding practices among slum-dwelling women from Pune
3. To explore the association of utilization of maternal healthcare services ante and postnatally with birth outcomes and infant growth
4. To examine the association of household food insecurity with maternal healthcare service utilization, birth outcomes and infant feeding and growth
5. To create a Social and Behavioural Change Communication (SBCC) module aimed at improving the uptake of maternal services and promoting complementary feeding of infants.

ELIGIBILITY:
Inclusion Criteria: Participant

1. is willing and able to give informed consent
2. has been residing in a slum for a minimum of 3 years
3. is aged between 18 to 49 years
4. has a child or children less than 2 years of age

Exclusion Criteria:

1. She is unwilling to consent to participate in the study
2. The age of her child or children is greater than 2 years.
3. The mother or child have any congenital / chronic conditions

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The study deals with assessment of utilization of maternal healthcare services
Study Population: Subjects will be recruited by house-to-house survey in two major slums currently serviced by the Research Institute in Pune city
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2025-03-07 (Actual); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of women who consumed at least 100 Iron Folic Acid tablets | Through study completion, an average of 1 year
  Percentage of women who consumed at least 100 Iron Folic Acid tablets
Percentage of women who consumed deworming tablets at least once during pregnancy | Through study completion, an average of 1 year
  Percentage of women who consumed deworming tablets at least once during pregnancy
Percentage of women who underwent delivery preparedness | Through study completion, an average of 1 year
  Percentage of women who underwent delivery preparedness
Percentage of women with knowledge of key danger signs during pregnancy | Through study completion, an average of 1 year
  Percentage of women with knowledge of key danger signs during pregnancy such as vaginal bleeding, severe headaches
Percentage of women who delivered at institution | Through study completion, an average of 1 year
  Percentage of women who delivered at institution
Percentage of women who stayed at a facility for at least 24 hours post-delivery | Through study completion, an average of 1 year
  Percentage of women who stayed at a facility for at least 24 hours post-delivery
Percentage of women who received post-natal care within a week of delivery | Through study completion, an average of 1 year
  Percentage of women who received post-natal care within a week of delivery
Percentage of women who availed at least three Antenatal Care (ANC) visits | Through study completion, an average of 1 year
  Percentage of women who availed at least three Antenatal Care (ANC) visits
Percentage of women who had contact with ASHA worker during pregnancy | Through study completion, an average of 1 year
  Percentage of women who had contact with Accredited Social Health Activist (ASHA) worker during pregnancy

SECONDARY OUTCOMES:
Association of demographic characteristics and household food insecurity scores with the indicators of utilization of healthcare services | Through study completion, an average of 1 year
  The association of demographic characteristics such as age of the participant, education of participant and her husband, occupation of participant and her husband, socio-economic status of the family, gender of the infant and household food insecurity scores will be investigated with each indicator of utilization of maternal healthcare service.

OTHER OUTCOMES:
Correlation of indicators of utilization of healthcare services with birth outcomes | Through study completion, an average of 1 year
  Correlation of the indicators of utilization of healthcare services with birth outcomes such as 1. gestational age at birth - preterm or term birth 2. birth weight - low birth weight or appropriate birth weight 3. gestational size - small for gestational age / appropriate for gestational age 4. Neonatal complications
Correlation of indicators of utilization of healthcare services with infant growth | Through study completion, an average of 1 year
  Correlation of the indicators of utilization of healthcare services with infant growth parameters such as 1. body weight 2. length 3. mid-upper arm circumference

CONTACTS AND LOCATIONS:
Overall Officials: Rubina M Mandlik, PhD, Principal Investigator — Hirabai Cowasji Jehangir Medical Research Institute
Locations (1):
- Hirabai Cowasji Jehangir Medical Research Institute, Pune, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No